CLINICAL TRIAL: NCT03063619
Title: A Randomized, Double-Blind, Placebo-Controlled Study of 4-hydroxytamoxifen Topical Gel in Women With Mammographically Dense Breast
Brief Title: Afimoxifene in Reducing the Risk of Breast Cancer in Women With Mammographically Dense Breast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-0328; NCI-2017-00244 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00034 (CTRP (Clinical Trial Reporting Program)); 2017-0328 (Other: MD Anderson Cancer Center); MDA2016-07-02 (Other: DCP); N01CN00034 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-02-24 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Mammographically Dense Breast
MeSH Terms: interventions — afimoxifene; 4,17 beta-dihydroxy-4-androstene-3-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (placebo) (Placebo Comparator): Patients apply placebo gel topically to each breast QD for up to 52 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Questionnaire Administration
- Arm B (afimoxifene) (Experimental): Patients apply afimoxifene gel topically to each breast QD for up to 52 weeks.
  Interventions: Drug: Afimoxifene; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Afimoxifene — Applied topically
  Other Names: 4-Hydroxy-Tamoxifen; 4-Hydroxytamoxifen; 4-OHT
  Arms: Arm B (afimoxifene)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Applied topically
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm A (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well afimoxifene works in reducing the risk of breast cancer in women with mammographically dense breast. Estrogen can cause the growth of breast cancer cells. Hormone therapy using afimoxifene may fight breast cancer by blocking the use of estrogen by the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate and compare the percent change in mammographic breast density (using Cumulus software) from baseline to month 12 in women applying 4mg afimoxifene (4-hydroxytamoxifen [4-OHT]) gel per breast versus placebo.

SECONDARY OBJECTIVES:

I. To compare the Cumulus versus (vs.) Volpara breast density measurement methods to estimate percent change in mammographic breast density from baseline to month 12 in women applying 4mg of 4-OHT gel per breast vs. placebo.

II. To compare the percentage of women who underwent a change in Breast Imaging Reporting and Data System (BIRADS) category, comparing pre-and post- treatment measurements, for recipients of active agent versus placebo.

III. To estimate percentage of women with >= 10% absolute decrease in quantitative mammographic density percentage between baseline and 12 months, comparing between treated group 4mg per breast 4-OHT gel to placebo.

IV. To describe symptoms assessed by breast cancer prevention trial (BCPT) eight symptom scale (BESS) questionnaire and laboratory toxicity assessment (factor VIII [F VIII], Von Willebrand [vWB] factor, sex hormone-binding globulin [SHBG], lipid profile).

V. To evaluate serum measurements of 4-OHT and related metabolite levels and factors related to tamoxifen exposures, such as insulin-like growth factor (IGF) pathway members, C-reactive protein (CRP), estradiol.

VI. To evaluate tissue biomarkers (among women undergoing optional pre- and post-treatment biopsies): terminal duct lobular unit (TDLU) involution; collagen structural changes; SETER/PR index: estrogen related transcription, Ki-67, COX-2, p16, CD68.

VII. To examine whether any reductions in mammographic density seen after 1 year of 4-OHT vs. placebo gel application persist at 24 months, one year after gel application has stopped.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients apply placebo gel topically to each breast once daily (QD) for up to 52 weeks.

ARM B: Patients apply afimoxifene gel topically to each breast QD for up to 52 weeks.

After completion of study treatment, patients are followed up at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Women age 40-69 years, or less than 40 years if 5-year breast cancer Gail risk is ≥ 1.66%.
* Mammographically dense breast (heterogeneously dense [C] or extremely dense [D], based on American College of Radiology [ACR] BIRADS fifth edition classification or heterogeneously dense [3] or extremely dense [4], based on ACR BIRADS fourth edition classification) in either breast
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* White blood cells >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 × institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits
* Participant must have a gynecology examination within the last 3 years, with no atypical hyperplasia and no cancer
* Premenopausal women taking non hormonal intra-uterine device (IUD) birth control method will be eligible, if they have been on the same IUD for at least 3 months prior to enrollment and plan to continue using the same method throughout the study
* Women of child-bearing potential must agree to use a reliable nonhormonal contraceptive method during the study and for 2 months after completing study medications; reliable nonhormonal methods of contraception include barrier contraception and an intra-uterine device (IUD); Note: women who had tubal ligation or had a partner who had undergone a vasectomy (and are monogamous) are eligible for the study and are not required to use barrier contraception
* If the participant is of childbearing potential, she must have a documented negative urine pregnancy test within 7 days prior to randomization
* Willingness to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the duration of the study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 4-OHT gel
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, thromboembolic disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant, or had given birth, or nursed at any time during the last 12 months
* Women with a previous history of invasive breast cancer or bilateral ductal carcinoma in situ (DCIS) or current untreated DCIS; women with a history of cancer within the last 3 years, except for non-melanoma skin cancer; women with unilateral DCIS (with or without radiation therapy) are eligible as long as they have an unaffected breast
* Prior bilateral breast surgery (mastectomy, segmental mastectomy, or breast augmentation surgery including breast implants or breast reductions)
* Women with "mosaic mammographic screening views", i.e., whose larger breast size precludes being imaged within a single mammographic screening view
* Women with active liver disease, abnormal uterine bleeding, or prior diagnosis of endometrial hyperplasia
* Prior use of selective estrogen receptor modulators (SERMS) and aromatase inhibitors (AIs) for prevention or therapy
* Skin lesions on the breast that disrupt the stratum corneum (e.g., eczema, ulceration)
* Treatment with any investigational drug or investigational biologic within 30 days of initiating study treatment or during the study

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 194 participants have been accrued, 158 randomized, 78 and 80 in 4-OHT gel and placebo, respectively.
Pre-assignment Details: Eleven participants withdrew consent, 19 ineligible, 6 other reasons (denied insurance, lost to follow-up, logistics).
Groups:
- 4-OHT Gel: Participants apply 4-OHT Gel topically to each breast QD for up to 52 weeks.
  4-OHT Gel: Applied topically
- Placebo: Participants apply Placebo gel topically to each breast QD for up to 52 weeks.
  Placebo: Applied topically
Period: Overall Study
Arm/Group | 4-OHT Gel | Placebo
Started | 78 | 80
Baseline | 78 | 80
Month 12 | 67 | 65
Month 24 | 56 | 55
Completed | 67 | 65
Not Completed | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-OHT Gel | Placebo | Total
Number analyzed (Participants) | 78 | 80 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 57 | 122
  >=65 years | 13 | 23 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 80 | 158
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 12 | 16
  Not Hispanic or Latino | 70 | 64 | 134
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 63 | 66 | 129
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 80 | 158

OUTCOME MEASURES:

1. Primary Outcome: Mammographic Breast Density Using Cumulus Software
Description: To determine change of mammographic breast density using Cumulus software. Cumulus is a semi-automated computerized measure of dense area that uses reader-based thresholds to define the breast edge and regions of density on a digital or digitized mammogram. Each pixel within the breast area between the skin line and pectoral muscle is segmented into either fat or fibro glandular tissue; this defines the cut-off point.
Time Frame: Baseline to Month 12
Population: Mammographic breast density data are available in a total of 133 participants, two without baseline data, six without month-12 data and two with 12-month mammograms beyond 18 months therefore are not considered evaluable for Month 12 evaluation. Therefore, a total of 123 participants are evaluable for the primary endpoint, 61 in 4-OHT and 62 in Placebo.
Measure: Mean (Standard Deviation); unit: Percent Change in Breast Density
Arm/Group | 4-OHT Gel | Placebo
Number analyzed (Participants) | 61 | 62
Percent Change in Breast Density
  Craniocaudal View (CC view) | -6.30 (9.11) | -5.77 (11.24)
  Mediolateral Oblique View (MLO view) | -2.81 (6.74) | -5.43 (9.08)

2. Secondary Outcome: Mammographic Breast Density Using Volpara Software
Description: To determine change of mammographic breast density using Volpara software. Volpara software uses a combination of x-ray physics and machine learning to generate an accurate volumetric measure of breast composition.
Time Frame: Baseline to Month 12
Population: A total of 59 participants have been evaluated for breast density at either baseline or month 12 or both by Volpara data, however 23 in 4-OHT and 24 in Placebo by CC view, and 25 in 4-OHT and 24 in Placebo by MLO view are evaluable for percent change in mammographic breast density.
Measure: Mean (Standard Deviation); unit: Percent Change in Breast Density
Arm/Group | 4-OHT Gel | Placebo
Number analyzed (Participants) | 32 | 27
Percent Change in Breast Density
  Craniocaudal View (CC view): number analyzed (Participants) | 23 | 24
  Craniocaudal View (CC view) | -1.31 (1.87) | -0.85 (2.35)
  Mediolateral Oblique View (MLO view): number analyzed (Participants) | 25 | 24
  Mediolateral Oblique View (MLO view) | -0.92 (4.26) | -0.30 (4.60)

3. Secondary Outcome: 4-OHT Plasma Levels
Description: To evaluate plasma measurements of 4-OHT levels, Z-4-OH-Tamoxifen.
Time Frame: Baseline to Month 12
Population: A total of 59 and 57 participants in 4-OHT and Placebo arms, respectively, have Month 12 measures on 4-OHT in plasma. All baseline measures are Below Qualification Limit (BQL).
Measure: Number; unit: participants
Arm/Group | 4-OHT Gel | Placebo
Number analyzed (Participants) | 59 | 57
participants
  Below Qualification Limit (BQL) at 12 months | 42 | 57
  Greater than BQL at 12 months | 17 | 0

4. Secondary Outcome: 4-OHT Tissue Levels
Description: To evaluate tissue measurements of 4-OHT levels, Z-4-OH-Tamoxifen
Time Frame: Baseline to Month 12
Population: A total of 12 and 18 participants in 4-OHT and Placebo arms, respectively, have Month 12 measures on 4-OHT in tissue. All baseline measures are Below Qualification Limit (BQL).
Measure: Number; unit: participants
Arm/Group | 4-OHT Gel | Placebo
Number analyzed (Participants) | 12 | 18
participants
  Below Qualification Limit (BQL) | 2 | 18
  Greater than BQL | 10 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Arm/Group | 4-OHT Gel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/80
Serious Adverse Events (participants affected / at risk) | 3/78 | 5/80
Other Adverse Events (participants affected / at risk) | 51/78 | 56/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4-OHT Gel (N=78) | Placebo (N=80)
Acute Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Perianal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Automobile Accident/Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Right Breast IDC/Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Breast Cancer/Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4-OHT Gel (N=78) | Placebo (N=80)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 2 (2) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspareunia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Entercolitis Infections (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2)
Fecal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 13 (13) | 16 (16)
Headache (Nervous system disorders) | 11 (11) | 8 (8)
Hot flashes (Vascular disorders) | 13 (13) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Irritability (General disorders) | 1 (1) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Olfactory nerve disorder (Nervous system disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Pain in extremity (General disorders) | 3 (3) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 3 (3)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Photosensitivity (General disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1)
Sore throat (Infections and infestations) | 0 (0) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Toothache (General disorders) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine obstruction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Dryness (Reproductive system and breast disorders) | 1 (1) | 4 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Weight gain (Investigations) | 6 (6) | 4 (4)
Weight loss (Investigations) | 3 (3) | 0 (0)
Wound Complication (Immune system disorders) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Breast Pain (Reproductive system and breast disorders) | 7 (7) | 7 (7)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03063619/Prot_SAP_000.pdf